CLINICAL TRIAL: NCT00773968
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once Monthly Administration of Subcutaneous C.E.R.A. for the Maintenance of Haemoglobin Levels in Pre-Dialysis Patients With Chronic Renal Anaemia
Brief Title: A Study of Monthly Subcutaneous Continuous Erythropoietin Receptor Activator (CERA) in Predialysis Participants With Chronic Renal Anemia
Acronym: ORION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21439; 2008-003173-40 (EudraCT Number)
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Methoxy Polyethylene Glycol-Epoetin Beta (Experimental): Participants will receive methoxy polyethylene glycol-epoetin beta once monthly by subcutaneous (SC) injection for 28 weeks.
  Interventions: Drug: Methoxy Polyethylene Glycol-Epoetin Beta

INTERVENTIONS:
Drug: Methoxy Polyethylene Glycol-Epoetin Beta — 120, 200 or 360 micrograms every 4 weeks by subcutaneous injection.
  Other Names: CERA

SUMMARY:
This single arm study will assess the long term maintenance of hemoglobin (Hb) levels, safety and tolerability of once monthly subcutaneous methoxy polyethylene glycol-epoetin beta (CERA) in predialysis participants with chronic renal anemia. Participants currently receiving subcutaneous darbopoetin alfa maintenance treatment will receive subcutaneous methoxy polyethylene glycol-epoetin beta for a maximum of 32 weeks at a starting dose of 120, 200 or 360 micrograms every 4 weeks according to the dose of darbopoetin alfa administered in Week -1. Subsequent doses will be adjusted to maintain hemoglobin levels within the target range of 10 to 12 grams per deciliter (g/dL).

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal anemia;
* Continuous subcutaneous maintenance darbopoetin alfa treatment during previous month;
* Hb concentration between 10 and 12 g/dL;
* Adequate iron status.

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months;
* Significant acute or chronic bleeding, such as overt gastrointestinal bleeding;
* Poorly controlled hypertension requiring hospitalization or interruption of darbopoetin alfa treatment in the previous 6 months;
* Active malignant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- Italy (34):
  - Barletta, Apulia
  - Molfetta (Ba), Apulia
  - Putignano, Apulia
  - Caserta, Campania
  - Eboli, Campania
  - Napoli, Campania
  - Nola, Campania
  - Solofra, Campania
  - Tivoli, Campania
  - Bologna, Emilia-Romagna
  - Pordenone, Friuli Venezia Giulia
  - Albano Laziale, Lazio
  - Civita Castellana, Lazio
  - Viterbo, Lazio
  - Savona, Liguria
  - Cinisello Balsamo, Lombardy
  - Cremona, Lombardy
  - Mantova, Lombardy
  - Monza, Lombardy
  - Pavia, Lombardy
  - S Fermo Della Battaglia, Lombardy
  - Varese, Lombardy
  - Campobasso, Molise
  - Alessandria, Piedmont
  - Chivasso, Piedmont
  - Catania, Sicily
  - Erice, Sicily
  - Messina, Sicily
  - Palermo, Sicily
  - Ancona, The Marches
  - Pesaro, The Marches
  - Lido di Camaiore, Tuscany
  - Pistoia, Tuscany
  - Siena, Tuscany

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants received methoxy polyethylene glycol-epoetin beta (also known as continuous erythropoietin receptor activator [CERA]) once monthly by subcutaneous (SC) injection, for 28 weeks. The initial dose of methoxy polyethylene glycol-epoetin beta was 120 or 200 or 360 micrograms (µg) if the last weekly dose of previous erythropoietin stimulating agent (ESA) (darbepoetin alfa) was less than (<) 40 µg or 40-80 µg or greater than (>) 80 µg, respectively. The doses were adjusted according to individual participant's hemoglobin (Hb) value.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Started | 140
Treated | 111
Completed | 95
Not Completed | 45
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Failure to Return | 2
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 11
Not completed — Screen Failure | 17
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who entered the study and received at least one dose of methoxy polyethylene glycol-epoetin beta.
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants received methoxy polyethylene glycol-epoetin beta once monthly by SC injection, for 28 weeks. The initial dose of methoxy polyethylene glycol-epoetin beta was 120 or 200 or 360 µg if the last weekly dose of previous ESA (darbepoetin alfa) was <40 µg or 40-80 µg or >80 µg, respectively. The doses were adjusted according to individual participant's Hb value.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Their Mean Hb Concentration Within Plus/Minus (±) 1 Grams Per Deciliter (g/dL) of the Reference Range and Between 10.0 and 12.0 g/dL During Efficacy Evaluation Period (EEP)
Description: The reference Hb was defined as the average Hb concentration calculated on the basis of all Hb assessments taken at Weeks -4, -2, and 0 (before the first dose administration).
Time Frame: EEP: Weeks 17 to 28
Population: Per protocol population included all participants who received at least one dose of methoxy polyethylene glycol-epoetin beta and for whom the data for at least one follow-up variable were available and were without any major protocol violation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 41
percentage of participants | 65.85 [49.41 to 79.92]

2. Secondary Outcome: Change in Hb Concentrations Between EEP and Stability Verification Period (SVP)
Description: Hb concentrations during SVP were the reference Hb concentrations. For each assessment period (SVP and EEP) the average Hb concentration was calculated on the basis of all Hb assessments taken during the assessment period. Change in average Hb concentration from reference range (SVP) was calculated.
Time Frame: SVP: Week -4 to Week 0; EEP: Weeks 17 to 28
Population: Per protocol population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 41
g/dL | 0.27 (0.73)

3. Secondary Outcome: Percentage of Participants Maintaining Hb Concentrations Within the Range of 10.0 to 12.0 g/dL Throughout EEP
Time Frame: EEP: Weeks 17 to 28
Population: Per protocol population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 41
percentage of participants | 73.17 [57.06 to 85.78]

4. Secondary Outcome: Median Time Spent in the Hb Range of 10.0 to 12.0 g/dL During the EEP
Time Frame: EEP: Weeks 17 to 28
Population: Per protocol population.
Measure: Median (Full Range); unit: days
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 41
days | 57.0 [0.0 to 86.0]

5. Secondary Outcome: Percentage of Participants Requiring Any Dose Adjustment During Dose Titration Period (DTP) and EEP
Description: The methoxy polyethylene glycol-epoetin beta dose adjustment (dose increase or decrease) was required: if a single Hb concentration was either greater than or equal to (≥) 13 g/dL or less than or equal to (≤) 9 g/dL; if the difference of 2 consecutive Hb concentrations was ≥2 g/dL; when the values of scheduled Hb assessments on the days of drug administration and on the previous study visit were both out of range of 10.5 to 11.5 g/dL and the difference between the reference value (average Hb concentration calculated on the basis of all Hb assessments taken at Weeks -4, -2, and 0) and the most recent value was >1 g/dL; and when the values of scheduled Hb assessments on the days of drug administration and on the previous study visit were both out of range of 10 to 12 g/dL. Dose adjustment could be made at any time at the discretion of the clinician if clinically warranted.
Time Frame: DTP: Weeks 1 to 16; EEP: Weeks 17 to 28
Population: Per protocol population.
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 41
percentage of participants
  DTP: Dose Increase Only | 17.1
  DTP: Dose Decrease Only | 39.0
  DTP: Both Dose Increase and Decrease | 22.0
  EEP: Dose Increase Only | 31.7
  EEP: Dose Decrease Only | 9.8
  EEP: Both Dose Increase and Decrease | 9.8

6. Secondary Outcome: Percentage of Participants Who Required Red Blood Cell Transfusions
Time Frame: Weeks 1 to 28
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 111
percentage of participants | 0.9

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: Safety population.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 10/111
Other Adverse Events (participants affected / at risk) | 14/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=111)
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Transaminases increased (Investigations) | 1
Renal impairment (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hospitalisation (Surgical and medical procedures) | 1
Extremity necrosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=111)
Renal impairment (Renal and urinary disorders) | 6
Hypertension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.